CLINICAL TRIAL: NCT01932151
Title: Terlipressin and Albumin in Patients With Type-1 Hepatorenal Syndrome Associated With Sepsis
Brief Title: Treatment of Type-1 Hepatorenal Syndrome Associated With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Pere Gines, Chairman, Liver Unit, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIN-TER-2010-01
Record Dates: First submitted 2013-08-14; First posted 2013-08-30 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Hepatorenal Syndrome
Keywords: type-1 HRS; active bacterial infections; terlipressin and albumin; kidney function
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Terlipressin; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Terlipressin and albumin (Other): Single-group study (Type-1 Hepatorenal Syndrome Associated With Active Infections) Terlipressin was initially given at a dose of 1 mg/4h as an intravenous bolus for 2 days. If at day 3 serum creatinine had decreased at least 25% of the pretreatment values, the dose of terlipressin was not modified. In the remaining patients, the dose was increased up to a maximum of 2 mg/4h. Terlipressin was given until serum creatinine had decreased below 1.5 mg/dL (133 µmol/L) or for a maximum of 14 days.
  Interventions: Drug: Terlipressin and albumin

INTERVENTIONS:
Drug: Terlipressin and albumin — Single-group study (Type-1 Hepatorenal Syndrome Associated With Active Infections) Terlipressin was initially given at a dose of 1 mg/4h as an intravenous bolus for 2 days. If at day 3 serum creatinine had decreased at least 25% of the pretreatment values, the dose of terlipressin was not modified. In the remaining patients, the dose was increased up to a maximum of 2 mg/4h. Terlipressin was given until serum creatinine had decreased below 1.5 mg/dL (133 µmol/L) or for a maximum of 14 days.
  In addition to terlipressin, all patients received albumin at a dose of 1g per kg body weight during the first 24 hours, followed by 40g daily,targeted to obtain a central venous pressure (CVP) between 10 and 15 cm of water.
  Other Names: - Glypressyn, Ferring SA, Saint-Prex, Switzerland.; - Albúmina Humana Grífols, Grífols , Barcelona, Spain.

SUMMARY:
Type 1 Hepatorenal syndrome (type-1 HRS) is a severe complication of patients with advanced cirrhosis characterized by marked renal failure and is associated with a very poor prognosis. Type-1 HRS is often precipitated by a bacterial infection, though it may occur spontaneously. It has been demonstrated that vasoconstrictor agents plus albumin are effective in the reversal of the renal failure. A large number of studies have shown that terlipressin improves renal function in patients with type 1 HRS; treatment is effective in 50-75% of patients approximately. Currently there are no specific studies about the treatment of type-1 HRS with ongoing infections.

DETAILED DESCRIPTION:
All consecutive patients with cirrhosis hospitalized with an infection or who developed an infection during hospitalization for an acute decompensation of the disease in four university hospitals.

Criteria for inclusion were: 1/ cirrhosis as diagnosed by liver biopsy or a combination of clinical, biochemical, ultrasonographic, and/or endoscopic findings; 2/ age between 18 and 80 years; 3/ presence of sepsis, as defined by infection and signs of Systemic Inflammatory Response Syndrome; and 4/ occurrence of type-1 HRS during the infection, as defined by standard diagnostic criteria. Exclusion criteria were: 1/ hepatocellular carcinoma outside the Milan criteria; 2/ any severe extrahepatic condition, including cardiovascular, neurological, and organic kidney diseases; 3/ septic or hypovolemic shock; 4/ terminal condition (death expected in less than 48 hours); and 5/ lack of informed consent.

Aim: A proof of concept study to evaluate whether treatment with terlipressin and albumin in the course of an infection associated with type-1 HRS is effective and safe.

ELIGIBILITY:
Inclusion criteria:

* Cirrhosis as diagnosed by liver biopsy or a combination of clinical, biochemical, ultrasonographic, and/or endoscopic findings.
* Age between 18 and 85 years.
* Presence of sepsis, as defined by active infection, and signs of Systemic Inflammatory Response Syndrome.
* Occurrence of type-1 HRS during the infection, as defined by standard diagnostic criteria.

Exclusion criteria:

* Hepatocellular carcinoma outside the Milan criteria.
* Any severe extrahepatic condition, including cardiovascular, neurological, and organic kidney diseases.
* Septic or hypovolemic shock.
* Terminal condition (death expected in less than 48 hours).
* Lack of informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in serum creatinine values | baseline and 14 days

SECONDARY OUTCOMES:
changes in glomerular filtration rate | at 3 days and 14 days
Changes in arterial pressure | baseline to 14 days
changes in plasma renin activity | at 3 days and 14 days
changes in norepinephrine concentration | at 3 days and 14 days

OTHER OUTCOMES:
Presence of adverse effects | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, MD, Principal Investigator — Hospital Clinc of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain